CLINICAL TRIAL: NCT03049202
Title: BROnchoalveolar Investigations of Never-smokers With CHronic Obstructive Lung Disease From the Swedish CardioPulmonary bioImage Study
Brief Title: BROnchoalveolar Investigations of Never-smokers With Chronic Obstruction From the Swedish CardioPulmonary bioImage Study
Acronym: BRONCOSCAPIS
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Lund University (Other); Göteborg University (Other); Linkoeping University (Other Government); Uppsala University (Other); Umeå University (Other); Karolinska University Hospital (Other); Lund University Hospital (Other); Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other); Uppsala University Hospital (Other); University Hospital, Umeå (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Asa Wheelock, Associate professor, Karolinska Institutet
Other Study IDs: 2016/841-31/2
Record Dates: First submitted 2017-01-31; First posted 2017-02-09 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis; Airway Obstruction; Smoking, Tobacco; Gender
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Airway Obstruction; Tobacco Smoking; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Mouth wash, bronchoalveolar lavage (BAL) cells, BAL fluid, bronchial wash (BW) cells, BW fluid, bronchial biopsies, airway epithelial brushings, serum, plasma, blood cells, and urine are collected and stored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Never-smoker COPD participants: COPD patients with mild-to-moderate COPD (GOLD I-II) that have never smoked. Definition of never-smoker: Lifetime consumption of <100 cigarettes. No cigarettes the past 2 years.
- Ex-smoker COPD participants: COPD patients with mild-to-moderate COPD (GOLD I-II) that stopped smoking. Definition of smoking: > 10 pack years. Definition of ex-smoker: > 2 years since smoke cessation.
- Current-smoker COPD participants: COPD patients with mild-to-moderate COPD (GOLD I-II) that are currently smoking. Definition of smoking: > 10 pack years. Definition of current-smoker: > 10/cigarettes/dat the past 6 months.
- Current-smoker healthy controls: Current-smokers that are otherwise healthy, with normal lung function. Definition of smoking: > 10 pack years. Definition of current-smoker: > 10/cigarettes/dat the past 6 months.
- Never-smoker healthy controls: Healthy participants that have never smoked. Definition of never-smoker: Lifetime consumption of <100 cigarettes. No cigarettes the past 2 years.

SUMMARY:
Obstructive lung disease is an increasing global health problem of pandemic proportions, with COPD alone affecting >10% of the population. Smoking is the main and most well studies risk factor for developing COPD. However, chronic airway obstruction also in never-smoking populations has recently been recognized as an increasing health problem.

In the clinical segment (PI: Prof. C. Magnus Skold), 1000 subjects from the Swedish national SCAPIS study will be clinically well characterized in one of the six Swedish University Hospital Respiratory clinics (clinical site PIs: Anders Andersson, Leif Bjermer, Anders Blomberg, Christer Janson, Lennart Persson, Magnus Skold). This first screening includes all never-smokers with COPD identified in the SCAPIS study. A subset of 300 subjects from the groups of Healthy never-smokers, current-smokers with normal lung function, current-smokers with COPD, ex-smokers with COPD, and never-smokers with COPD will be selected for the Bronchoscopy segment, were sampling will be performed from a number of anatomical locations, including bronchial biopsies, airway epithelial brushings, and bronchoalveolar lavage. Serum, plasma, and urine samples will also be collected.

In the systems medicine segment (PI: Assoc. prof Asa M. Wheelock), alterations at the epigenetic, mRNA, microRNA, proteome, metabolome and microbiome level will be performed from multiple lung compartments (airway epithelium, alveolar macrophages, exosomes, and bronchoalveolar exudates). By means of biostatistics and bioinformatics approaches, specific mediators and molecular pathways critical in the pathological mechanisms of obstructive lung disease related to never-smoker disease phenotypes will be identified.

In the immunohistochemistry segment (PI: Prof. Jonas Erjefalt), a number of molecules of relevance for disease pathology will be investigated in bronchial biopsies collected from the 300 subjects in the Bronchoscopy segment.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an umbrella diagnosis defined by obstructive lung function impairments, and is likely to be caused by a multitude of etiologies including environmental exposures, genetic predispositions and developmental factors. Due to the heterogeneity of the disease, molecular and mechanistic sub-phenotyping of COPD represents an essential step to facilitate the development of relevant diagnostic and treatment options for this constantly growing patient group. In the BRONCHO-SCAPIS study, molecular sub-phenotypes of smoking-induced COPD are investigated. A particular focus relates to recent epidemiological indications of an increasing proportion of never-smokers developing the disease. The study encompasses profiling of mRNA, miRNA, proteomes, metabolomes and lipid mediators of from multiple lung compartments (airway epithelium, alveolar macrophages, exosomes, and bronchoalveolar exudates) using a range of 'omics platforms, in combination with extensive clinical phenotyping of early stage COPD patients, never-smokers, and smokers with normal lung function from both genders. The primary objective of the study is to identify molecular sub-phenotypes of never-smokers with COPD, specifically by correlating clinical phenotypes multi-molecular 'omics profiling from multiple lung compartments of early stage COPD patients compared to healthy and at-risk control populations. Secondary goals involve identification of subsets of prognostic/diagnostic biomarkers for classification of the defined subgroups, as well as relevant pharmaceutical targets.

ELIGIBILITY:
Inclusion Criteria:

* Spirometry of postbronchodilator forced expiratory volume in 1 second (FEV1) >50% of predicted level for all groups.
* Spirometry of postbronchodilator FEV1 >80% of predicted level and FEV1/FVC ratio >0.70 for Healthy control groups
* Spirometry of postbronchodilator FEV1/FVC ratio <0.70 for COPD groups.

Exclusion Criteria:

* Smoking (for never-smoker groups)
* Other lung diseases
* Received antibiotics in the 3 months prior to study entry
* Treatment with oral or inhaled glucocorticoids within past 3 months prior to study entry

Ages: 50 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The 1000 participants are recruited from the Swedish SCAPIS study, a cross sectional study screening 30,000 subjects across the six University Hospitals in Sweden, based on lung function criteria and questionnaire criteria collected during SCAPIS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | Measured at baseline
  Calculated as percent predicted based on the European Coal and Steel Community reference values
Emphysema, as shown on chest CT scan | Measured at baseline
  Based on lung densities < (-950) Hounsfield units (HU)
Airway wall thickness on chest CT scan | Measured at baseline
  Based on lung densities in the range of (-750) - (-900) HU
COPD status (COPD participants versus control group participants) based on GOLD criteria | Measured at baseline
  Calculated using, post-bronchodilator values defined as meeting the criteria based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) of a fixed FEV1/forced vital capacity (FVC) ratio < 0.7
COPD status (COPD participants versus control group participants) based on GLI criteria | Measured at baseline
  Calculated using, post-bronchodilator values defined as meeting the Global Lung Initiative (GLI) ratio of FEV1/FVC below of lowest limit of normal z-score < (-1.64)

SECONDARY OUTCOMES:
Molecular phenotypes of never-smoker COPD group(s) as compared to control groups | Measured at baseline
  mRNA, miRNA, proteomes, lipidomes and metabolomes will be quantified from airway exudates (BAL fluid), BAL cells, and airway epithelium (bronchial brushings)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Skold, MD, PhD, Principal Investigator — Karolinska Institutet /Karolinska University Hospital
Locations (6):
- Sweden (6):
  - Karolinska Institutet/Karolinska University Hospital Solna, Stockholm, Sverige
  - Göteborg University / Sahlgrenska University Hospital, Gothenburg
  - Linköping Unversity /Linköping University Hospital, Linköping
  - Lund University / Lund University Hospital, Lund
  - Umeå University / Umeå University Hospital, Umeå
  - Uppsala University / Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No